CLINICAL TRIAL: NCT03509974
Title: Early Experience of a New Implant System for Bone Conduction Hearing in the Pediatric Population
Acronym: OSIA Pediatric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM5706
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Results first posted 2021-02-01 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Unilateral Mixed Conductive and Sensorineural Hearing Loss (Diagnosis); Sensorineural Hearing Loss, Unilateral With Normal Hearing on the Contralateral Side
MeSH Terms: conditions — Hearing Loss, Sensorineural; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bone Anchored Hearing Device (OSIA) (Experimental): All subjects will receive the Bone Anchored Hearing Device (OSIA)
  Interventions: Device: Osseointegrated Steady State Implant

INTERVENTIONS:
Device: Osseointegrated Steady State Implant — Bone anchored, bone conduction hearing system
  Other Names: Bone anchored, bone conduction hearing system

SUMMARY:
To study the initial experience with implanting and fitting a new Bone Conduction system in pediatric patient population with conductive, mixed or single-sided deafness.

DETAILED DESCRIPTION:
Experimental: Bone-conduction hearing device The bone-conduction hearing device Osia system allows a direct bone-conduction through an osseointegrated implant. A magnet allows the external Sound Processor to be placed in the correct position over the implanted system including an inner magnet.

Device: Osia System An external Sound Processor captures and digitize the sound which is transferred to the internal implant where it is converted to an electrical signal. The electrical signal is further transferred as a vibration through an osseointegrated implant to the mastoid bone and eventually to the cochlea

ELIGIBILITY:
Inclusion Criteria: Individuals 5 through 18 years of age will be eligible for inclusion in the investigation if all of the criteria below are met:

Conductive or mixed hearing loss in the ear to be implanted. Bone conduction thresholds with pure-tone average (PTA4; mean of 0.5, 1, 2, and 4 kHz) of less than or equal to 55 dB HL.

Subject does not benefit from or will not wear a conventional hearing aid.

Note: Candidates may include individuals seeking new implantation unilaterally (in one ear) or bilaterally (both ears) as well as individuals already implanted with a bone-anchored device seeking a second-side implant.

OR

Single-sided sensorineural deafness who is a candidate for Baha surgery. Air conduction thresholds with a pure-tone average (PTA4; mean of 0.5, 1, 2, and 3 kHz) of less that equal to 20 dB HL in the good ear.

Subject does not benefit from or will not wear a conventional hearing aid

Exclusion Criteria:

Uncontrolled diabetes as judged by the investigator. Subject who has received radiotherapy in the area of implantation, or such radiotherapy is planned during the study period.

Current use of ototoxic drugs. Condition that could jeopardize osseointegration and/or wound healing or condition that may have an impact on the outcome of the investigation as judged by the investigator.

Insufficient bone quality and quantity for implantation of a BI300 Implant, as determined by the surgeon.

Unable to follow investigational procedures. Participation in another clinical investigation with pharmaceutical and/or device

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bone Anchored Hearing Device (OSIA)
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bone Anchored Hearing Device (OSIA)
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Type of Hearing Loss [Count of Participants; unit: Participants]
  Conductive | 9
  Mixed Conductive | 2
  Single-Sided-Deafness | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Type and Severity of Adverse Events in the Pediatric Population Implanted With the Osia System
Description: Number, Type and Severity of Adverse Events will be tabulated and summarized.
Time Frame: Surgery to 12 months post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Anchored Hearing Device (OSIA)
Number analyzed (Participants) | 14
Participants
  Not Serious - Ingrown hair near incision | 1
  Not Serious - Red incision site with pus leaking | 1
  Not Serious - Patient bumped magnet site in shower, pain and swelling | 1
  Serious - Skin flap measurement >10mm prevented device connectio/activiation | 1
  Not Serious - Pain and swelling at the tip of mastoid | 1
  Not Serious - magnetitis and soe discomfort with pin skin | 1
  Not Serious - right swelling at the tip of the mastoid | 1
  Not Serious - Left side facial swelling at post-operative site | 1
  Not Serious - Redness at magnet site | 1
  Not Serious - some discomfort following surgery | 1
  Not Serious - Pain and swelling at surgical sight | 1
  Not Serious - Post-operative nausea and vomitting | 1
  Not Serious - swelling post surgery | 1
  Not Serious - Sensitivity post surgery | 1
  Not Serious - discomfort post surgery for one week | 1

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Bone Anchored Hearing Device (OSIA)
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Anchored Hearing Device (OSIA) (N=14)
Prevention of Device Connection/Activation (Ear and labyrinth disorders) | 1 (1) — Skin flap easurement greater than 10mm prevented device connection/activation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Anchored Hearing Device (OSIA) (N=14)
Ingrown hair near incision site (Injury, poisoning and procedural complications) | 1 (1)
Red incision site with some pus leaking (Injury, poisoning and procedural complications) | 1 (1)
Pain and swelling at magnet site (Product Issues) | 1 (1) — Patient bumped magnet site leadig to pain and swelling
Pain and swelling at the tip of mastoid (Product Issues) | 1 (1)
Magnetitis and discomfort (Product Issues) | 1 (1) — Very mild magnetitis causing pink skin
Right swelling at the tip of the mastoid (Product Issues) | 1 (1)
Left-side facial swelling at post-operation (Injury, poisoning and procedural complications) | 1 (1)
Redness at magnet site (Product Issues) | 1 (1)
Some discomfort following surgery (Injury, poisoning and procedural complications) | 1 (1)
Pain and swelling at surgical site (Injury, poisoning and procedural complications) | 1 (1)
Post-operation nausea and vomitting (Injury, poisoning and procedural complications) | 1 (1)
Swelling post surgery (Injury, poisoning and procedural complications) | 1 (1)
Sensitivity post surgery (Injury, poisoning and procedural complications) | 1 (1)
Discomfort post-surgery (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators and Team at Sick Kids preparing a publication for peer review with sponsor coordination.

DOCUMENTS (1):
  • Study Protocol (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT03509974/Prot_000.pdf